CLINICAL TRIAL: NCT02694952
Title: Randomized, Double-blind, Non-inferiority Trial of Two Antivenoms for the Treatment of Snakebite With Envenoming
Brief Title: Non-inferiority Trial of Two Snake Antivenoms in CAR (PAVES)
Acronym: PAVES
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ministry of Health in country did not authorized the conduct of the study
Sponsor: Epicentre (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPICENTRE CAR 2016
Record Dates: First submitted 2016-02-17; First posted 2016-03-01 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Snake Bites
MeSH Terms: conditions — Snake Bites

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FAV-Africa (Active Comparator): FAV-Africa infusion at enrollment, and then at two and six hours after enrollment, if necessary. To be given as unblinded rescue dose at twelve hours if fourth dose of antivenom necessary.
  Interventions: Biological: FAV-Africa
- EchiTabPlus-ICP (Experimental): EchiTabPlus-ICP infusion at enrollment, and then at two and six hours after enrollment, if necessary.
  Interventions: Biological: EchiTabPlus-ICP

INTERVENTIONS:
Biological: FAV-Africa — Polyspecific antivenom immunoglobulin F(ab)'2 fragments of equine origin manufactured by Sanofi Pasteur, S.A., Lyon, France. Per undiluted 1 ml, the multivalent serum contains ≥25 times the LD50 for mice exposed to venom of Bitis gabonica, Bitis arietans, Echis leucogaster, Echis ocellatus, Naja haje, Dendroaspis polylepis, Dendroaspis viridis, and Dendroaspis jamesoni, as well as ≥20 times the LD50 for mice exposed to venom of Naja melanoleuca and Naja nigricollis.
  Arms: FAV-Africa
Biological: EchiTabPlus-ICP — Polyspecific antivenom immunoglobulin of equine origin manufactured by the Clodomiro Picado Institute, San Jose, Costa Rica. Each 10 ml of undiluted antivenom contains enough antibody fragments to neutralize 30 mg of Echis ocellatus venom, 20 mg of Bitis arietans venom and 5 mg of Naga nigricollis venom.
  Arms: EchiTabPlus-ICP

SUMMARY:
Interventional, individually randomized, double (e.g. investigator and participant) blinded, parallel two-arm, non-inferiority trial to assess the efficacy of EchiTabPlus-ICP compared to FAV-Africa for the treatment of snakebite with envenoming.

DETAILED DESCRIPTION:
The study is designed as a randomized, double-blind, non-inferiority trial among patients suffering envenoming following snakebite in Paoua, Central African Republic. The primary aim of the study is to assess the non-inferiority of EchiTabPlus-ICP compared to FAV-Africa, at preventing a composite primary endpoint consisting of death from any cause, need for blood transfusion or need for a third dose of antivenom.

A total of 196 patients will be individually randomized in a 1:1 ratio to receive FAV-Africa or EchiTabPlus-ICP.

The first dose of intervention antivenom will be administered at study enrollment, and the need for further doses will be judged by clinical exam and the 20 minute WBCT, following the protocol. All other necessary medical care will be provided as per routine in the Paoua Prefectural Hospital. Study followup and surveillance for adverse events and serious adverse events will continue until 28 days after the initial dose of antivenom.

Unique identification numbers will be allocated by an individual independent of the study team using a computer-generated random number list using permuted blocks of random sizes. Block sizes will not be disclosed to reduce predictability of the random sequence and ensure allocation concealment. The Site Principal Investigator who will oversee randomization will be given a set of sequentially numbered silver coated booklets. The Site Principal Investigator will be instructed to assign the next sequential randomization code noted in the booklet to each eligible participant as (s)he is enrolled.

Study antivenoms will be prepared by the unblinded study pharmacist, and will be provided to the clinical staff in identical presentations. Group assignment will remain concealed from study personnel, investigators, and participants for the entire study period. The Data and Safety Monitoring Board (DSMB) will also be masked to the group assignment. The DSMB will remain masked unless otherwise deemed necessary by the DSMB members for any safety related issues. Investigators conducting the final analysis will remain masked to the group assignment until the end of the analysis.

ELIGIBILITY:
Inclusion Criteria:

* present within 72 hours of snakebite
* have signs and symptoms of grade 2 envenoming (oedema beyond the elbows or knees, bleeding at site of bite, bleeding from the gums or hematuria) or grade 3 envenoming (oedema to the shoulders or hips, or serious bleeding - epistaxis, hemoptysis, gastrointestinal bleeding)
* lack of coagulation of blood at 20 minutes in a dry vacutainer tube (abnormal 20 minute WBCT)

Exclusion Criteria:

* known allergy to horses or heterologous proteins of equine origins
* pregnancy
* have received antivenom since the snakebite

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03 (Estimated); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of patients needing a third dose of antivenom, needing a blood transfusion, or dying | 28 days after enrolment

SECONDARY OUTCOMES:
Death from any cause | 28 days after enrolment
Need for blood transfusion | Will be evaluated at 2, 6, 12, and 24 hours after enrolment and at hospital discharge
Need for third dose of antivenom | Will be evaluated at 2, 6, 12, and 24 hours after enrolment and at hospital discharge
Normalization of coagulopathy as measured by the 20 minute whole blood clotting test | Will be evaluated at 2, 6, 12, and 24 hours after enrolment
  Using 20 min whole blood clotting test

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Grais, PhD, Study Director — Epicentre

IPD SHARING:
Plan to Share IPD: No